CLINICAL TRIAL: NCT00774306
Title: The Effects of Antiepileptic Drugs on Serum Lipids and Inflammation in Patients With Subarachnoid Hemorrhage
Brief Title: Antiepileptic Drugs and Vascular Risk Markers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study no longer consistent with current clinical practice
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23NS058669 (NIH); 1K23NS058669 (NIH)
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Subarachnoid Hemorrhage
Keywords: vascular risk; lipid fractions; lipoprotein(a); C-reactive protein; subarachnoid hemorrhage; antiepileptic drug; randomized; seizure; cholesterol
MeSH Terms: conditions — Subarachnoid Hemorrhage; Seizures | interventions — Phenytoin; fosphenytoin; Valproic Acid; Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Participants randomized to Group 1 will receive phenytoin (PHT) at 5 mg/kg/day in 2 divided doses.
  Interventions: Drug: phenytoin
- 2 (Active Comparator): Participants randomized to Group 2 will receive valproate (VPA) at 15 mg/kg/day in 3 divided doses or in a once-daily extended release formulation.
  Interventions: Drug: valproate
- 3 (Active Comparator): Participants randomized to Group 3 will receive levetiracetam (LEV) 1000-1500 mg/day in 2 divided doses.
  Interventions: Drug: levetiracetam
- 4 (No Intervention): Participants randomized to Group 4 will receive no drug intervention.

INTERVENTIONS:
Drug: phenytoin — Phenytoin is a anti-seizure medication. Participants will receive phenytoin (PHT) at 5 mg/kg/day in 2 divided doses.
  Other Names: Dilantin, Cerebyx (a phenytoin pro-drug)
  Arms: 1
Drug: valproate — Valproate is an anti-seizure medication. Participants will receive valproate (VPA) at 15 mg/kg/day in 3 divided doses.
  Other Names: Depakote, Depacon
  Arms: 2
Drug: levetiracetam — Levetiracetam is an anti-seizure medication. Participants will receive levetiracetam (LEV) 1000-1500 mg/day in 2 divided doses.
  Other Names: Keppra
  Arms: 3

SUMMARY:
The purpose of this study is to determine if certain seizure medications raise levels of cholesterol and other blood components which could increase the risk of heart attacks and strokes.

DETAILED DESCRIPTION:
There is some evidence that certain seizure medicines may raise levels of cholesterol and other blood components which could increase the risk of heart attacks and strokes, however, more research is needed. Individuals with acute subarachnoid hemorrhage traditionally are treated with seizure medicines, but it is not clear which one is best, or if any such medication is necessary at all.

This study is intended to find out if certain seizure medications raise levels of cholesterol and other blood components which could lead to an increased risk of heart attacks and strokes.

In this study, 200 people with acute subarachnoid hemorrhage will be randomized to treatment with one of three different seizure medicines-phenytoin, valproate, or levetiracetam-or to receive no seizure medication at all. In each participant, cholesterol and other blood markers that relate to heart attack and stroke risk will be measured shortly after hospital admission and again 8 weeks later. At the 8-week point most participants will have their seizure medication discontinued, and the same blood tests will be repeated.

Information from this study could lead to changes in how seizure medications are prescribed both in the subarachnoid hemorrhage population and in other people who are prone to seizures.

ELIGIBILITY:
Inclusion Criteria:

* Acute subarachnoid hemorrhage, Hunt-Hess Grades I-IV
* Within 48 hours of admission

Exclusion Criteria:

* Grade V subarachnoid hemorrhage
* Being treated with a lipid-lowering agent
* Contraindication to phenytoin, valproate, or levetiracetam (e.g. history of allergy to one of these agents)
* Contraindication to receiving no antiepileptic drug treatment (e.g. history of pre-existing epilepsy, seizure activity on admission EEG)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Mintzer, MD, Principal Investigator — Assistant Professor of Neurology, Jefferson Comprehensive Epilepsy Center

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenytoin: Participants randomized to Group 1 will receive phenytoin (PHT) at 5 mg/kg/day in 2 divided doses.
  phenytoin: Phenytoin is a anti-seizure medication. Participants will receive phenytoin (PHT) at 5 mg/kg/day in 2 divided doses. They will be maintained on it throughout the study period. Daily dose will be adjusted to maintain levels in the standard therapeutic range of 10-20 mg/dL. Upon discharge, they will remain on the drug in oral form until follow-up with the principal investigator 6 weeks later.
  x
  x
- Valproate: Participants randomized to Group 2 will receive valproate (VPA) at 15 mg/kg/day in 3 divided doses or in a once-daily extended release formulation.
  valproate: Valproate is an anti-seizure medication. Participants will receive valproate (VPA) at 15 mg/kg/day in 3 divided doses.
- Levetiracetam: Participants randomized to Group 3 will receive levetiracetam (LEV) 1000-1500 mg/day in 2 divided doses.
  levetiracetam: Levetiracetam is an anti-seizure medication. Participants will receive levetiracetam (LEV) 1000-1500 mg/day in 2 divided doses.
- No Anticonvulsant: Participants randomized to Group 4 will receive no drug intervention.
Period: Overall Study
Arm/Group | Phenytoin | Valproate | Levetiracetam | No Anticonvulsant
Started | 24 | 5 | 16 | 7
Completed | 6 | 3 | 8 | 2
Not Completed | 18 | 2 | 8 | 5
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 6 | 1 | 1 | 0
Not completed — Lost to Follow-up | 6 | 0 | 4 | 5
Not completed — Death | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phenytoin: Participants randomized to Group 1 will receive phenytoin (PHT) at 5 mg/kg/day in 2 divided doses.
  phenytoin: Phenytoin is a anti-seizure medication. Participants will receive phenytoin (PHT) at 5 mg/kg/day in 2 divided doses.
- Total: Total of all reporting groups
Arm/Group | Phenytoin | Valproate | Levetiracetam | No Anticonvulsant | Total
Number analyzed (Participants) | 24 | 5 | 16 | 7 | 52
Age, Continuous [Median (Full Range); unit: years] | 48.5 [31 to 71] | 46 [26 to 62] | 51 [30 to 71] | 49 [44 to 75] | 48 [26 to 75]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 5 | 14 | 5 | 46
  >=65 years | 2 | 0 | 2 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 10 | 6 | 34
  Male | 10 | 1 | 6 | 1 | 18
Region of Enrollment [Number; unit: participants]
  United States | 24 | 5 | 16 | 7 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Cholesterol, Non-HDL Cholesterol, HDL Cholesterol, Lipoprotein(a), and C-reactive Protein From Baseline to Second Draw and Third Draw in Each of the 4 Study Arms
Time Frame: 8 weeks, 16 weeks
Groups:
- Phenytoin: Participants randomized to Group 1 will receive phenytoin (PHT) at 5 mg/kg/day in 2 divided doses.
  phenytoin: Phenytoin is a anti-seizure medication. Participants will receive phenytoin (PHT) at 5 mg/kg/day in 2 divided doses. They will be maintained on it throughout the study period.
  x
  x
Arm/Group | Phenytoin | Valproate | Levetiracetam | No Anticonvulsant
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Incidence of Acute Seizures, Incidence of Late Seizures, Overall Neurologic Function (as Measured by Modified Rankin Scale Scores)
Time Frame: 8 weeks, 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Phenytoin | Valproate | Levetiracetam | No Anticonvulsant
Serious Adverse Events (participants affected / at risk) | 4/24 | 1/5 | 4/16 | 3/7
Other Adverse Events (participants affected / at risk) | 0/24 | 1/5 | 0/16 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phenytoin (N=24) | Valproate (N=5) | Levetiracetam (N=16) | No Anticonvulsant (N=7)
vasospasm (Nervous system disorders) | 1 | 1 | 2 | 1
deep venous thrombosis (Vascular disorders) | 1 | 0 | 1 | 0
hydrocephalus (Nervous system disorders) | 1 | 0 | 1 | 0
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
drug fever (Immune system disorders) | 1 | 0 | 0 | 0
cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phenytoin (N=24) | Valproate (N=5) | Levetiracetam (N=16) | No Anticonvulsant (N=7)
urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Study terminated due to 1) change in clinical practice; 2) inadequate recruitment and follow-up.

Number of pts providing full data was <15% of goal. Because of this, any analysis of data was considered futile, and no analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No